CLINICAL TRIAL: NCT03778918
Title: The Comparison Between That Expression Pattern and Disease Activity of Variable Biomarkers in Inflammatory Bowel Disease Patients and General Control Group. Multicenter, Prospective Study
Brief Title: The Comparison Between the Biomarkers in Inflammatory Bowel Disease Patients and General Control Group
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bo-In Lee (Other)
Collaborators: Incheon St.Mary's Hospital (Other); St Vincent's Hospital (Other); Daejeon St. Mary's hospital (Other)
Responsible Party: Sponsor-Investigator, Bo-In Lee, Professor, MD, PhD., Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: XC18TEDI0027
Record Dates: First submitted 2018-12-09; First posted 2018-12-19 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome
Keywords: REG3 alpha; IBD; biomarker; ulcerative colitis; serum calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Blood, Biopsy tissue, Stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inflammatory bowel disease: inflammatory bowel disease such as Ulcerative colitis and Crohn's disease
  Interventions: Other: inflammatory bowel disease; Other: IBS or Normal Control
- IBS or Normal Control: irritable bowel syndrome patients normal patients
  Interventions: Other: inflammatory bowel disease; Other: IBS or Normal Control

INTERVENTIONS:
Other: inflammatory bowel disease — blood based biomarkers in IBD such as REG3 alpha, serum calprotectin and hs-CRP
Other: IBS or Normal Control — blood based biomarker compared normal control with IBD

SUMMARY:
The aims of this study is to investigate a blood-based biomarker that can replace endoscopy in patients with inflammatory bowel disease. For this purpose, blood sample of patients wiht inflammatory bowel disease (ulcerative colitis, Crohn 's disease) was collected at the same time the endoscopy is performed, stored after centrifugation, and analyzed accordingly. Selected biomarkers from the blood sample were investigated to compare those of patients with inflammatory bowel disease and those of general controls. Males and females over the age of 19 participated in the study and are excluded if they have chronic kidney disease or blood clotting disease. The outcome is a find of a blood-based biomarker that best reflects a disease activity.

DETAILED DESCRIPTION:
Inflammatory bowel disease refers to chronic inflammation of the unknown origin that occurs in the intestine. It usually refers to ulcerative colitis and Crohn's disease, which are idiopathic inflammatory bowel diseases. While it had been known to be a common disease in the western world, in recent decades the incidence of ulcerative colitis and Crohn's disease has rapidly increased in Korea as well. Endoscopic examination is a gold standard in order to determine the activity of inflammatory bowel disease, but it is hardly performed due to the cost and time of a test. Therefore, it is necessary to find a blood-based biomarker that replaces endoscopy. The objective of the study is to identify a new inflammatory marker that replaces endoscopy by comparing blood samples of patients with inflammatory bowel disease with those of general controls.

ELIGIBILITY:
Inclusion Criteria:

* people who receive colonoscopy
* people who sign the consent
* having inflammatory bowel disease (ulcerative colitis, Crohn's Dz.) and irritable bowel syndrome

Exclusion Criteria:

* those aged over 75 years
* the disabled
* pregnant women
* chronic renal diseases (CLcr <50ml/min)
* blood coagulopathy (PT INR > 1.5, aPTT > 45 seconds, or platelet count < 50,000/mm)
* people who refuse to sign the consent

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: inflammatory bowel disease (ulcerative colitis, Crohn's Dz.) irritable bowel syndrome normal control
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
measurement of blood-based biomarkers to predict disease activity 1 | within 12 weeks of the blood sampling
  REG3 alpha (ng/mL)
measurement of blood-based biomarkers to predict disease activity 2 | within 12 weeks of the blood sampling
  hs-CRP (mg/dL)
measurement of blood-based biomarkers to predict disease activity 3 | within 12 weeks of the blood sampling
  serum calprotectin (ng/mL)

SECONDARY OUTCOMES:
Age (years) | at the time of study enrolled
  age at the time of study enrolled
Gender (M/F) | at the time of study enrolled
  male of female
disease duration (months) | at the time of study enrolled
  duration of disease
disease onset (years) | at the time of study enrolled
  age at which the disease begins

CONTACTS AND LOCATIONS:
Overall Officials: Bo-In Lee, MD. Ph.D., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Division of Gastroenterology; Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darnaud M, Dos Santos A, Gonzalez P, Augui S, Lacoste C, Desterke C, De Hertogh G, Valentino E, Braun E, Zheng J, Boisgard R, Neut C, Dubuquoy L, Chiappini F, Samuel D, Lepage P, Guerrieri F, Dore J, Brechot C, Moniaux N, Faivre J. Enteric Delivery of Regenerating Family Member 3 alpha Alters the Intestinal Microbiota and Controls Inflammation in Mice With Colitis. Gastroenterology. 2018 Mar;154(4):1009-1023.e14. doi: 10.1053/j.gastro.2017.11.003. Epub 2017 Nov 11. PMID 29133078
- [Background] Greuter T, Lang S, Holler E, Hawkey CJ, Rogler G, Biedermann L; ASTIC trial group. Serum REG3alpha and C-Reactive Protein Levels in Crohn's Disease Patients Undergoing Immunoablation and Autologous Hemopoetic Stem Cell Transplantation in the ASTIC Trial. Digestion. 2015;92(2):83-9. doi: 10.1159/000437300. Epub 2015 Aug 1. PMID 26278889
- [Background] Harris AC, Levine JE, Ferrara JL. Have we made progress in the treatment of GVHD? Best Pract Res Clin Haematol. 2012 Dec;25(4):473-8. doi: 10.1016/j.beha.2012.10.010. Epub 2012 Oct 25. PMID 23200544